CLINICAL TRIAL: NCT06636864
Title: Effect of Intrathecal Morphine on Quality of Recovery After Laparoscopic Colorectal Cancer Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, RenChun Lai, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-FXY-302
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Colorectal Cancer Surgery
Keywords: Laparoscopic colorectal cancer surgery; QoR-15; Intrathecal morphine
MeSH Terms: interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal morphine group (Experimental): Before induction of anesthesia, the experimental group received intrathecal morphine in the lumbar segment (L3/4).For our preliminary clinical application, the intrathecal morphine was 3ug/kg
  Interventions: Procedure: Intrathecal morphine; Procedure: TAPB
- Normal saline group (Active Comparator): Before anesthesia induction, the control group received intrathecal injection of normal saline.
  Interventions: Procedure: Intrathecal saline injection; Procedure: TAPB

INTERVENTIONS:
Procedure: Intrathecal morphine — The patient was asked to lie on the side, the needle insertion point was located under the guidance of color ultrasound, and after local anesthesia, the needle was inserted into the subarachnoid space at the puncture point and morphine was injected.
  Arms: Intrathecal morphine group
Procedure: Intrathecal saline injection — After the patient was asked to lie on his side, the injection point was determined under the guidance of color ultrasound. After local anesthesia, the needle was injected into the subarachnoid space and then normal saline was injected.
  Arms: Normal saline group
Procedure: TAPB — The patient was in a supine position. The rectus muscle was confirmed to be warping under the guidance of color photography, and the needle was injected with bupivacaine liposomes

SUMMARY:
Colorectal cancer is the second most common tumor in women and the third most common tumor in men, accounting for approximately 10% of tumors diagnosed and tumor-related deaths worldwide each year. Laparoscopic resection has become the standard of colorectal cancer surgery, and its main advantages are to shorten the length of hospital stay, reduce postoperative pain, and accelerate patient recovery. However, it has been reported that about 49% of patients undergoing laparoscopic colorectal cancer surgery still have moderate to severe postoperative pain. The insertion of abdominal drainage tube will increase the degree of postoperative pain, especially when patients take deep breaths, exercise or cough, which will increase the demand for postoperative opioids and reduce the quality of postoperative recovery. How to further reduce the postoperative pain of patients, reduce the dosage of opioids, shorten the length of hospital stay, promote the rapid recovery of patients and improve patient satisfaction are our concerns. Intrathecal morphine can provide a good analgesic effect on visceral pain. At present, intrathecal morphine has become a new method of postoperative analgesia, which is used in thoracic, abdominal and obstetrics and gynecology operations. The objective of this study was to investigate the effect of intrathecal morphine on the quality of recovery after laparoscopic colon cancer surgery.

DETAILED DESCRIPTION:
Colorectal cancer is the second most common tumor in women and the third most common tumor in men, accounting for approximately 10% of tumors diagnosed and tumor-related deaths worldwide each year. Laparoscopic resection has become the standard of colorectal cancer surgery, and its main advantages are to shorten the length of hospital stay, reduce postoperative pain, and accelerate patient recovery. However, it has been reported that about 49% of patients undergoing laparoscopic colorectal cancer surgery still have moderate to severe postoperative pain. The insertion of abdominal drainage tube will increase the degree of postoperative pain, especially when patients take deep breaths, exercise or cough, which will increase the demand for postoperative opioids and reduce the quality of postoperative recovery. How to further reduce the postoperative pain of patients, reduce the dosage of opioids, shorten the length of hospital stay, promote the rapid recovery of patients and improve patient satisfaction are our concerns.

The anesthesia scheme was endotracheal intubation general anesthesia combined with bupivacaine liposome plane block of transverse abdominal muscle, experimental group combined with intrathecal morphine, control group injected with intrathecal saline. Heart rate, electrocardiogram, pulse oxygen saturation, noninvasive blood pressure, and end-expiratory partial carbon dioxide pressure (ETCO2) were routinely monitored after entry. Before anesthesia induction, the experimental group received lumbar morphine (L3/4). Based on the literature and our previous clinical application, the intrathecal morphine was 3ug/kg. Control group received intrathecal injection of normal saline. General anesthesia was induced by intravenous injection of dexmedetomidine (0.5ug/kg), cyclopofol (0.4mg/kg), remifentanil (TCI4ng/ml) and rocuronium (0.6mg/kg), followed by tracheal intubation. Bupivacaine liposome plane block of transverse abdominal muscle was performed in both groups, bupivacaine liposome injection (20ml: 266mg) was diluted with 0.9% sodium chloride solution from 20ml to 40ml, and 10ml diluent solution was injected into the left and right abdominal subcostoal approach and lateral approach under ultrasound guidance. Anesthesia was maintained with 1-1.3MAC desflurane, remifentanil, sufentanil, cis-atracurium, and vasoactive agents as needed. Intraoperative opioid dosage was recorded. Patients in both groups received intravenous controlled analgesia, 150mg morphine with 0.9% sodium chloride solution to 150ml intravenous analgesia pump. The background dose is 0ml/h, the single patient-controlled analgesia dose is 1ml, and the locking time is 6 minutes to manage fulminant pain. When adverse events such as hypotension occur, appropriate accelerated fluid rehydration is given while makingWith vasoactive drugs, the nurse (who did not participate in the study) was asked to reduce the parameters of the intravenous analgesic pump to 1/2 of the original, and if the symptoms persisted, the analgesic pump was turned off and the study was terminated. The main outcome was QoR15 score 24 hours after operation.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic colorectal cancer surgery under tracheal intubation and general anesthesia is intended
* Agreed to use intravaginal morphine injection and bupivacaine liposomal plane block of transversal muscle after surgery
* ASA Grade I - III
* Over 18 years of age

Exclusion Criteria:

* Preoperative accident or subjective refusal of surgery
* Nervous system dysfunction
* Contraindications to intraspinal anesthesia
* Preoperative opioid use history
* Patients with abnormal preoperative pain and pain score (NRS) >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
QoR15 score at 24 hours after surgery | Day 1 after surgery

SECONDARY OUTCOMES:
QoR15 scores 48 and 72 hours after surgery | Day 2and 3 after surgery
Morphine consumption equivalent 24, 48, 72 hours after surgery | Day 1，2and 3 after surgery
Rest and cough NRS scores in PACU after surgery | 30 minutes after surgery
NRS scores at rest, deep breathing, activity, and cough 24, 48, and 72 hours after surgery | Day 1，2and 3 after surgery
Intraoperative opioid dosage | in surgery
First postoperative exhaust time | up to one week
The first time to get out of bed after surgery | up to one week
Supplement the amount of analgesic drugs 24, 48 and 72 hours after surgery | Day 1，2and 3 after surgery
Adverse events (dizziness, headache, nausea and vomiting, pruritus, hypotension) 24, 48, 72 hours after surgery | Day 1，2and 3 after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng L, Lu Y, Lu X, You L, Yu C, Lai J, Xu M, Xie M, Xiao Y, Lai R. Intrathecal Morphine for Enhanced Recovery After Laparoscopic Colorectal Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 Dec 23:e255699. doi: 10.1001/jamasurg.2025.5699. Online ahead of print. PMID 41433024